CLINICAL TRIAL: NCT06181578
Title: Efficacy and Safety Study of Adjunctive Ganglionated Plexus Ablation in Patients With Persistent Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: Ganglion Plexus Ablation in Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ning Zhou (Other)
Responsible Party: Sponsor-Investigator, Ning Zhou, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zn101516
Record Dates: First submitted 2023-11-29; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Atrial Fibrillation, Persistent; Ganglionated Plexi; Catheter Ablation
Keywords: persistent atrial fibrillation; catheter ablation; ganglionated plexus; high-frequency stimulation; autonomic nervous system; treatment outcome; randomized controlled trial
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study employs a single-blind design, where the research staff is aware of the patient's group assignment, but the patients themselves are unaware of their group allocation. This approach is implemented to minimize potential subjective bias. The research staff will make efforts to maintain blinding during interactions with the patients to ensure objectivity in data collection and outcome assessment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP Ablation Group (Experimental): Participants in this group will undergo a combined intervention, including standard ablation (pulmonary vein isolation and linear ablation) and additional ablation targeting the autonomic ganglionated plexus (GP).
  Interventions: Procedure: ganglionated plexus ablation
- Standard Ablation Group (No Intervention): Participants in this group will undergo standard ablation treatment, which includes pulmonary vein isolation (PVI) and linear ablation.

INTERVENTIONS:
Procedure: ganglionated plexus ablation — This intervention involves the targeted ablation of ganglionated plexus sites, specifically focusing on the left superior ganglionated plexus (LSGP), left inferior ganglionated plexus (LIGP), right anterior ganglionated plexus (RAGP), and right inferior ganglionated plexus (RIGP).
  Arms: GP Ablation Group

SUMMARY:
This study aims to investigate the long-term efficacy and safety of incorporating ganglionated plexus ablation into radiofrequency ablation strategies for persistent atrial fibrillation.

DETAILED DESCRIPTION:
1. Study Design:

   The study employs a parallel-group design with a 1:1 randomization ratio. Eligible patients meeting the specified criteria will be randomly assigned to either the conventional ablation group (pulmonary vein isolation + linear ablation) or the intervention group receiving additional ganglionated plexus ablation.
2. Intervention:

   Control Group: Conventional ablation (pulmonary vein isolation + linear ablation) Intervention Group: Conventional ablation + ganglionated plexus ablation (left superior, left inferior, right anterior, and right inferior ganglionated plexi)
3. Randomization and Sequence Generation:

To ensure randomness and comparability, a computer-generated random sequence will be utilized. Specific steps include:

* Pre-matching the numbers 1-50 with 50 random numbers.
* Allocating each random number equally to 2 groups, with the assigned numbers representing the order of patient enrollment.
* Performing the above steps using R.

  5. Data Collection: Baseline data, including demographics, medical history, and laboratory parameters, will be collected at the start. Intraoperative electrophysiological and ablation-related parameters, as well as postoperative adverse events, will be documented. Follow-up data will include postoperative survival, quality of life (assessed using the Atrial Fibrillation Effect on Quality-of-Life questionnaire), dynamic electrocardiogram recordings, recurrence of atrial fibrillation or other arrhythmias, rehospitalization for arrhythmia, and medication usage.

  6. Endpoints:
* Primary Endpoints:

Recurrence of atrial tachyarrhythmias; Echocardiographic parameters; Procedure-related adverse events

* Secondary Endpoints:

Atrial fibrillation burden; Radiofrequency ablation time; Patient postoperative quality of life; Healthcare resource utilization

The trial's initiation date will be documented, and all procedures will be conducted at the Cardiovascular Department of Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, China. The study will adhere to ethical guidelines and regulations, and informed consent will be obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years, regardless of gender.
* Patients confirmed by electrocardiogram or clinically diagnosed with persistent atrial fibrillation.
* Individuals scheduled to undergo atrial fibrillation catheter ablation.
* Willing to participate in the study and voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients with a history of prior atrial fibrillation ablation surgery.
* Left ventricular ejection fraction (LVEF) less than 35%.
* Left atrial anterior-posterior diameter greater than 50mm on echocardiography.
* Presence of contraindications for atrial fibrillation ablation, such as the presence of clear thrombus in the left atrium detected preoperatively.
* Patients with second-degree (Type II) or third-degree atrioventricular block.
* Individuals with significant congenital heart defects (such as atrial septal defects or severe pulmonary vein stenosis, excluding unclosed foramen ovale).
* Patients with implanted artificial valves.
* Diagnosed with hypertrophic cardiomyopathy, chronic obstructive pulmonary disease, or myxoma.
* Untreated or uncontrolled hyperthyroidism or hypothyroidism.
* Patients with active systemic infections.
* Individuals with a significant bleeding tendency or those undergoing active blood dialysis due to renal failure.
* Patients who have experienced myocardial infarction within the last 3 months or undergone any cardiac intervention/open-heart surgery.
* Presence of clear contraindications for interventional procedures, as determined by the investigator.
* Pregnant or lactating women, or those planning pregnancy during the study period.
* Participation in other drug or medical device clinical trials within the last 3 months.
* Patients deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Atrial Tachycardia and Time to Recurrence | 91 to 365 days post-catheter ablation.
  The first occurrence of sustained atrial arrhythmias (excluding atrial premature beats) lasting ≥30 seconds recorded between 91 to 365 days post-catheter ablation, including atrial fibrillation and atrial flutter, etc.
Left Atrial Dimensions | 1 to 365 days post-catheter ablation.
  Measurement of left atrial size, a key indicator of atrial remodeling, assessed as a primary outcome to evaluate the impact of the intervention on atrial structure.
Left Ventricular Ejection Fraction, LVEF | 1 to 365 days post-catheter ablation.
  Assessment of left ventricular ejection fraction as a primary outcome measure, providing crucial insights into post-intervention cardiac function and guiding the evaluation of the treatment's efficacy on overall heart performance.
Procedure-Related Adverse Events | 1 to 365 days post-catheter ablation.
  Occurrence of adverse events related to the procedure during the perioperative or follow-up period, including but not limited to death, myocardial infarction, cardiac tamponade, and stroke.

SECONDARY OUTCOMES:
Atrial Fibrillation Burden | 91 to 365 days post-catheter ablation.
  Quantification of the burden of atrial fibrillation episodes throughout the follow-up period.
Radiofrequency Ablation Time | Recorded during the catheter ablation procedure.
  Total duration of radiofrequency ablation during the procedure.
Patient's Postoperative Quality of Life | 1 to 365 days post-catheter ablation.
  Assessment using the Atrial Fibrillation Effect on Quality-of-Life (AFEQT) questionnaire, providing insights into the impact of the procedure on the patient's quality of life.
Costs of treatment | From patient admission to discharge, averaging a duration of 3 days.
  Including expenses associated with medical procedures, hospital stay, and additional healthcare resources. The treatment costs will be expressed as a relative ratio, calculated by dividing the treatment cost per patient by the mean treatment cost of the control group.

IPD SHARING:
Plan to Share IPD: No